CLINICAL TRIAL: NCT03772158
Title: A Randomized, Single-Dose, Four-Treatment Crossover Bioequivalence and Food Effect Study of Test Formulation of Cetirizine 10mg Chewable Tablets Versus Two Marketed Cetirizine 10mg Immediate Release Tablets.
Brief Title: Cetirizine Chewable Bioequivalence and Food Effect Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc., McNeil Consumer Healthcare Division (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CCSURA000499
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Allergy
Keywords: Bioequivalence study; Healthy volunteers; Cetirizine; Tablet
MeSH Terms: conditions — Hypersensitivity | interventions — Cetirizine

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-dose, four-treatment crossover bioequivalence and food effect study of Cetirizine Chewable Tablets versus ZYRTEC® Immediate Release (IR) Tablets (US reference) and REACTINE® IR Tablets (EU and Australian marketed reference product).
  The study will be conducted in two parts. Part 1 of the study will have a randomized, four way crossover study design in which 40 healthy subjects, ages 18 to 55 years, will be randomized to four sequences of Treatments A, B, D and E over consecutive periods. No less than approximately 40% of either gender will be represented in the study population. Part 2 of the study will assess a potential food effect in which all subjects will be administered Treatment C in the fifth period.
Who Masked: Outcomes Assessor
Masking Description: Blinding of the test and reference products to study subjects is not feasible, because the products are different dosage forms (chewable tablets and IR tablets) and administered in different ways (with or without water and fasted or fed). Personnel conducting the bioanalyses of samples will not know the treatment sequence. The randomization code will not be available to them until the analytical tables have been finalized and audited by the Algorithme Pharma (An Altasciences Company) Quality Assurance (QA) department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Treatment A (Experimental): Single dose of 10 mg cetirizine as a chewable tablet, administered orally after a 10-hour overnight fast and followed with 240 mL ambient water. Subjects will be instructed to chew the tablet completely before swallowing.
  Interventions: Drug: Cetirizine 10mg
- Treatment B (Experimental): Single dose of 10 mg cetirizine as a chewable tablet, administered orally after a 10-hour overnight fast without water. Subjects will be instructed to chew the tablet completely before swallowing.
  Interventions: Drug: Cetirizine 10mg
- Treatment C (Experimental): Single dose of 10 mg cetirizine as a chewable tablet, administered orally after a 10-hour overnight fast and 30 minutes after the start of the standard high-fat breakfast and followed with 240 mL ambient water. Subjects will be instructed to chew the tablet completely before swallowing.
  Interventions: Drug: Cetirizine 10mg
- Treatment D (Active Comparator): Single dose of currently marketed US 10 mg cetirizine as immediate release tablet (ZYRTEC®), administered orally after a 10-hour overnight fast and followed with 240 mL ambient water.
  Interventions: Drug: Cetirizine 10 mg
- Treatment E (Active Comparator): Single dose of currently marketed EU/Australian 10 mg cetirizine film coated tablet (REACTINE®) administered orally after a 10-hour overnight fast and followed with 240 mL ambient water.
  Interventions: Drug: Cetirizine 10 mg

INTERVENTIONS:
Drug: Cetirizine 10mg — Chewable tablet
  Other Names: Test product
  Arms: Treatment A; Treatment B; Treatment C
Drug: Cetirizine 10 mg — Immediate Release Tablet
  Other Names: ZYRTEC 10 mg
  Arms: Treatment D
Drug: Cetirizine 10 mg — Immediate Release Tablet
  Other Names: REACTINE 10 mg
  Arms: Treatment E

SUMMARY:
The purpose of this study is to determine and compare the amount of study drug that gets into your blood after the administration of each of the three formulations of cetirizine under different conditions. Another objective of this study is to evaluate the effect of food on the amount of study drug that gets into your blood after the administration of the investigational formulation. Other objectives of this study are to determine the sensory experience and ease of swallowing the investigational formulation, as well as to determine the safety of test and reference formulations of cetirizine.

DETAILED DESCRIPTION:
The purpose of this study is to establish bioequivalence of a cetirizine 10 mg chewable tablet manufactured at Johnson & Johnson Consumer Inc. (McNeil LLC) with two commercially marketed cetirizine 10 mg immediate release (IR) tablets (ZYRTEC®, US reference) and (Australian/EU reference), establish bioequivalence between the two commercial products (ZYRTEC®, US reference and REACTINE®, Australian/EU reference), and to evaluate the effect of food on bioavailability of the cetirizine 10 mg chewable tablet compared to the bioavailability of cetirizine 10 mg chewable tablet administrated with water only. In addition, subject's sensory experience and ease of swallowing of the test product will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subject between the ages of 18 and 55 years, inclusive. Health is defined as the absence of clinically relevant abnormalities as judged by the Investigator on the basis of a detailed medical history, physical examination, blood pressure, pulse rate measurements, 12-lead electrocardiogram (ECG), as well as clinical laboratory tests. The responsible Investigator may request additional investigations or analyses if necessary.
2. Non- or ex-tobacco user, being defined as someone who completely stopped smoking or using any form of tobacco or nicotine-containing product for at least 6 months before screening visit of this study.
3. For females: Postmenopausal state (i.e. at least 1 year without menses without an alternative medical condition prior to the first study drug administration) or premenopausal /perimenopausal state with an effective means of contraception (as defined in Section 10.5.5).
4. For males: No pregnant or lactating spouse or partner at screening and willingness to utilize an acceptable form of birth control with spouse or any potential partner during the study.
5. Body Mass Index (BMI) ≥ 18.5 and ≤ 30 kg/m2 with a total body weight >50 kg.
6. A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.
7. Is able to comprehend the requirements of the study (based upon clinical site personnel's assessment) and is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures specified within the protocol.

Exclusion Criteria:

1. Use of prescription or non-prescription medications within 5 half-lives before the first IP administration unless these are contraceptives or occasional use of other medications approved by the Investigator.
2. Use of any vitamins, dietary and herbal supplements within seven days before first dose of study drug.
3. History of any allergy or hypersensitivity (e.g. skin reaction, asthma, angioedema) to cetirizine or any excipients of the formulations.
4. If female: is pregnant, has a positive pregnancy test at screening or prior to the first study drug administration, or is planning to become pregnant during the duration of the study, and/or is breast-feeding.
5. Has a history of gastrointestinal surgery other than appendectomy.
6. Has hypertension, fluid retention, or heart disease either by history or by the medically qualified Investigator's medical judgment.
7. Currently suffering from asthma or has a medically significant history of asthma in the opinion of the investigator.
8. Has clinically significant renal or hepatic impairment; according to the medically qualified Investigator discretion.
9. Was treated with an investigational product within 28 days or within a period less than 5 times the drug's half-life, whichever is longer, preceding the first dose of study drug.
10. Preplanned surgical procedures during the study period as this may interfere with the conduct of the study.
11. History of alcoholism or substance abuse, as judged by the Investigator, within the past 6 months preceding this study.
12. Consumed alcohol beverage(s) within 48 hours preceding the first dose of study drug.
13. History of rare hereditary problems of galactose and/or lactose intolerance, lactase deficiency or glucose-galactose malabsorption.
14. Any history of tuberculosis.
15. Donation or loss of blood within 28 days prior to the first treatment visit if the estimated lost blood volume equaled or exceeded 50 mL.
16. Donation or loss of blood within 56 days prior to the first treatment visit if the estimated lost blood volume equaled or exceeded 500 mL.
17. Has any acute or chronic medical or psychiatric condition(s) that may increase the risk associated with study participation or IP administration or may interfere with the interpretation of study results and, in the judgment of the medically qualified Investigator, would make the subject inappropriate for entry into this study.
18. Relationship to persons involved directly in the conduct of the study (i.e., principal Investigator, sub-Investigators, study coordinators, other study personnel, employees or contractors of the sponsor or Johnson & Johnson subsidiaries, and the family of each).
19. Has any clinically important abnormal value for serum chemistry, hematology, or urinalysis at screening. Laboratory values will generally be within the normal ranges, although minor deviations in tests (except those explicitly specified in the inclusion criteria) that are not considered clinically important by the Investigator are acceptable.
20. Has a positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (anti-HCV).
21. Has a positive test for alcohol or drugs of abuse at screening or prior to the first study drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — No less than approximately 40% of either gender will be represented in the study population.
Enrollment: 40 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2019-02-03 (Actual)

PRIMARY OUTCOMES:
The maximum observed plasma concentration (Cmax) of cetirizine | At baseline, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 28 and 32 hours after the start of dose administration.
  The maximum observed plasma concentration.
The area under the plasma concentration versus time curves to the last measurable concentration (AUCt) | At baseline, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 28 and 32 hours after the start of dose administration.
  Area under the plasma concentration versus time curve from start of drug administration until last measurable concentration.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve extrapolated to infinity | At baseline, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 28 and 32 hours after the start of dose administration.
  Area under the plasma concentration-time curve extrapolated to infinity.
The time point at which the maximum concentration of cetirizine is observed (Tmax). | At baseline, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 28 and 32 hours after the start of dose administration.
  The time point at which the maximum concentration of cetirizine occurs.
The terminal elimination half-life (T1/2) of cetirizine in plasma | At baseline, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 28 and 32 hours after the start of dose administration.
  The time it takes for the cetirizine plasma concentration to fall to half of its original value.
The terminal elimination rate constant (lambda z) for cetirizine in plasma. | At baseline, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 28 and 32 hours after the start of dose administration.
  The rate at which the drug is removed from the body system.
To assess subject's sensory experience and ease of swallowing of the test product | Assessed one minute after dosing, and preferably completed within 15 minutes of dosing for treatments A, B and C
  A questionaire with 5 product sensory questions for study subjects to answer.
Number of patients with adverse events. | Approximately 3 months. From signed informed consent until 30 days after last treatment administration.
  An adverse event is any untoward medical occurrence in a subject after they have signed an informed consent for a trial involving an investigational product.
The extrapolated part of the area under the plasma concentration versus time curve of cetirizine | Extrapolated from 12 hours after start of drug administration until 48 hours
  The area under the plasma concentration versus time curve from 12 hours after start of drug administration until 48 hours after start of drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme (An altascience Company), Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: CSR synopsis for Bioequivalence Study. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSURA000499&attachmentIdentifier=b1bd7d49-7220-4c5f-8c78-555f34b49b1d&fileName=CSR_CCSURA000499_Section_2_Synopsis_Redacted.pdf&versionIdentifier=